CLINICAL TRIAL: NCT07102069
Title: Pharmacogenomic and Pharmacoepigenomic Studies of Antipsychotic Drugs in First-Episode Schizophrenia
Status: Completed | Type: Observational
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJAH2017-SCH-LJ
Record Dates: First submitted 2025-07-18; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cohort Study; Cognition; Biomarker
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will retain peripheral blood samples collected at baseline and follow-up visits. These samples will be stored at -80 °C for future DNA extraction, genotyping, and methylation analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- schizophrenic patients: In this trial, a total of 300 schizophrenia patients who were never treated with antipsychotic medications or other psychotropics were recruited from out- or in-patients in Tianjin Anding Hospital. There are no restrictions for the types of antipsychotics. The enrolled patients received assessments at the main visits (baseline, week8, week12,1-year,2-year,5-year).
- healthy control: 100 healthy subjects were matched to patients in age, sex, race, and education. They completed the same baseline assessment as the patients. what's more, part of the enrolled healthy group will receive an assessment at week8 follow-up.

SUMMARY:
This study aims to explore the objective markers concerning schizophrenia risk and functional outcome from multiple dimensions such as multi-omics including genomics, proteomics, metabolomics, electrophysiology, imaging, psychosocial, and cognition. In summary, based on this trial, the significant outcomes may effectively improve the accuracy of early warning and recognition in patients with schizophrenia, and provide clues for the study of new drug targets.

DETAILED DESCRIPTION:
This trial is a prospective, longitudinal observation clinical trial. In this trial, a total of 300 SZ patients who were never treated with antipsychotic medications or other psychotropics were recruited from out- or in-patients in Tianjin Anding Hospital. Patients received antipsychotic treatment at the discretion of their clinicians. The types of antipsychotics were not restricted. In this longitudinal study, all patients received clinical evaluation scales including the Positive and Negative Syndrome Scale (PANSS), and so on at the main visits (baseline, week8, week12, 1-year, 2-year, 5-year). Importantly, cognitive evaluation using the MATRICS Consensus Cognitive Battery (MCCB) and functional Magnetic Resonance Imaging (fMRI) imaging were collected only at five follow-ups（baseline，week8， 1-year， 2-year， 5-year）. Meanwhile, we also collect related measured factors by collecting a peripheral blood sample and electrophysiological index including Electroencephalogram (EEG) and Functional Near-Infrared Spectroscopy (fNIRS) at multiple time points (baseline, week8, week12, 1-year, 2-year,5-year). 100 healthy subjects were matched to patients in age, gender, race, and education. They completed the same baseline assessment as the patients. what's more, part of the enrolled healthy group will receive an assessment at week8 follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy population matched with gender, age, and educational level of case group;
* Han nationality;
* Sign informed consent.

Exclusion Criteria:

* Major physical and brain diseases;
* Any mental disorder in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV);
* Parents have a family history of mental illness in two lines and three generations;
* Currently taking psychoactive drugs;
* Refuse to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this trial, a total of 300 schizophrenia patients who were never treated with antipsychotic medications or other psychotropics were recruited. And the case group received assessments including clinical evaluation scales, collecting peripheral blood samples, and so on at the main visits (baseline, week8, week12,1-year,2-year,5-year). Importantly there are no restrictions on the types of antipsychotics. 100 healthy subjects considering age, gender, race, and years of education controls completed the same baseline assessment as the patients at baseline. what's more, part of the enrolled healthy group will receive an assessment at week8 follow-up.
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Changes of psychiatric symptoms | Baseline, week8, week12, 1year, 2year, 5year
  The psychiatric symptoms of schizophrenia were assessed in all enrolled patients using the Positive and Negative Syndrome Scale (PANSS). The PANSS is a 30-item clinician-rated scale yielding a total score ranging from 30 (least symptomatic) to 210 (symptomatic), where higher scores indicate more severe psychopathology. Trained raters administered the PANSS at multiple follow-up visits: baseline, Week 8, Week 12, 1 year, 2 years, and 5 years.
Changes of cognitive function | Baseline, week8, 1year, 2year, 5year
  All subjects received baseline cognitive evaluation using the MATRICS Consensus Cognitive Battery (MCCB). It involves seven cognitive areas: (1) Speed of Processing Information; (2) Attention and Vigilance Awareness; (3) Working Memory; (4): Verbal Learning; (5) Visual Learning; (6) Reasoning and Problem-Solving; (7) Social Cognition. The MCCB scoring program generates T-scores that are standardized and corrected for age and sex. A higher T score indicates better cognitive function. The cognitive composite is the standardized sum of the seven domains.

SECONDARY OUTCOMES:
Allelic Frequency of Target Single-Nucleotide Polymorphisms (SNPs) | Baseline
  We will quantify the allelic frequency of pre-specified SNPs using DNA extracted from peripheral blood. Results are reported as the percentage of each allele (%) at each locus.
Gene-Specific DNA Methylation Level | Baseline
  We will measure DNA methylation at CpG sites within candidate genes using bisulfite pyrosequencing. Results are reported as the percentage (%) of methylated cytosines at each interrogated site.
Changes of C-reactive protein (CRP) levels | Baseline, week8, week12
  Serum CRP will be quantitatively measured using an enzyme-linked immunosorbent assay. The results will be expressed as the absolute change in CRP concentration (mg/L) between the baseline value and the measured value, with higher values indicating more severe systemic inflammation.
Changes of interleukin-1β (IL-1β) levels | Baseline, week8, week12
  Serum IL-1β will be quantitatively measured using an enzyme-linked immunosorbent assay. The results will be expressed as the absolute change in CRP concentration (pg/mL) between the baseline value and the measured value, with higher values indicating more severe systemic inflammation.
Changes of interleukin-6 (IL-6) levels | Baseline, week8, week12
  Serum IL-6 will be quantitatively measured using an enzyme-linked immunosorbent assay. The results will be expressed as the absolute change in CRP concentration (pg/mL) between the baseline value and the measured value, with higher values indicating more severe systemic inflammation.
Changes of tumour necrosis factor-α (TNF-α) levels | Baseline, week8, week12
  Serum TNF-α will be quantitatively measured using an enzyme-linked immunosorbent assay. The results will be expressed as the absolute change in CRP concentration (μg/L) between the baseline value and the measured value, with higher values indicating more severe systemic inflammation.
Resting-State electroencephalography (EEG) Relative Power | Baseline
  Resting-state EEG will be recorded with 32-channel active electrodes at 1 kHz sampling. Relative power in the theta (4-8 Hz) and alpha (8-13 Hz) bands will be calculated using fast Fourier transform.
Functional near-infrared spectroscopy (fNIRS) | Baseline
  The fNIRS will be used to monitor oxygenated hemoglobin (HbO₂) and deoxygenated hemoglobin (Hb) in the bilateral prefrontal cortex during a working-memory task.
Resting-state functional magnetic resonance imaging (fMRI) | Baseline
  A single resting-state BOLD-fMRI scan will be acquired at baseline using a 3 T scanner (TR=2000 ms, TE=30 ms, voxel size=3 mm isotropic). Functional connectivity between the dorsolateral prefrontal cortex (seed) and the whole brain will be computed as Fisher-z transformed correlation coefficients. The outcome is the baseline connectivity strength expressed as z-score; higher positive z-scores indicate stronger connectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No